CLINICAL TRIAL: NCT05917964
Title: A Randomized, Two-period, Two-sequence Two-treatment Crossover Design Food Effect Study to Evaluate the Pharmacokinetic Profile of LP-168 Tablets in Healthy Subjects After Single Oral Administration Under Fasted and Fed Conditions
Brief Title: A Food Effect Study of LP-168 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LP-168-CN103
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (fasted-fed) (Experimental): Cohort A was administered once in Cycle 1 Day1 under fasted condition and once in Cycle 2 Day1 (i.e., Day8 after Cycle 1 administration) under fed condition for a total of 2 doses.
  Interventions: Drug: LP-168 tablet
- Cohort B (fed-fasted) (Experimental): Cohort B was administered once in Cycle 1 Day 1 under fed condition and once in Cycle 2 Day 1 (i.e., D8 after Cycle 1 administration) under fasted conditions for a total of 2 doses.
  Interventions: Drug: LP-168 tablet

INTERVENTIONS:
Drug: LP-168 tablet — LP-168 is a small molecule kinase inhibitor that is administered once daily via oral administration
  Other Names: NWP-775

SUMMARY:
This is a randomized, two-period, two-sequence two-treatment crossover design food effect study to evaluate the pharmacokinetic profile of LP-168 tablets in healthy subjects after single oral administration under fasted and fed conditions

DETAILED DESCRIPTION:
A total of 22 subjects from Cohort A and Cohort B, with a single sex ratio of not less than 1/3, will be included in this study. Each subject will undergo two cycles of self-crossover dosing, respectively. 4 days of PK sample collection and safety observation period will be conducted after the first dose for the first cycle, followed by the 4-day second cycle of PK sample collection and safety observation. The washout period between the 2 doses will be 7 days.

Subjects who voluntarily participate in the study and complete the informed consent process will be randomly assigned to the fasted-fed group (Cohort A) or the fed-fasted group (Cohort B) in a 1:1 ratio after completion of all screening visit examinations and after the investigator determines that all inclusion criteria are met and all exclusion criteria are not met. Cohort A was administered once in Cycle 1 Day1 under fasted condition and once in Cycle 2 Day1 (i.e., Day8 after Cycle 1 administration) under fed condition for a total of 2 doses; cohort B was administered once in Cycle 1 Day 1 under fed condition and once in Cycle 2 Day 1 (i.e., D8 after Cycle 1 administration) under fasted conditions for a total of 2 doses, both at a dose of 150 mg of LP-168 tablets.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have no history of serious digestive system, central nervous system, cardiovascular system, kidney, respiratory system, metabolism and endocrine, skeletal and muscular system, blood system disease and cancer
* Subjects (including partners) are willing to take effective contraception measures during study and within 3 months after last dose
* Male and female healthy subjects aged 18 to 55 years old
* Male subjects weigh ≥ 50 kg, and female subjects weigh ≥ 45 kg
* Subjects able to understand and comply with study requirements
* Willing to sign the informed consent

Exclusion Criteria:

* Abnormal vital signs, physical examination or laboratory tests with clinical significance
* Abnormal ECG or echocardiography with clinical significance
* Hepatitis B virus, Hepatitis C virus, HIV and syphilis test positive. COVID-19 DNA positive.
* Subjects who have taken any drugs or health care products within 14 or 28 days before administration the study drug
* Subjects who have consumed diets that may alter the activity of liver metabolic enzymes within 7 days before administration the study drug
* Subjects who have consumed tea or alcohol-containing food product within 24hrs before administration the study drug
* Subjects who have a history of dysphagia or condition may affect drug absorption, distribution, metabolism and excretion
* Female subjects are breastfeeding or pregnant
* Subjects who have a history of drug/ alcohol/ tobacco abuse
* Subjects who have had a blood donation or massive blood loss within three months before screening; or had surgery within six months before screening
* Subjects who have participated in other clinical trial within three months before screening
* Subjects have special dietary requirements or cannot tolerate a standard meal

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
PK Parameter AUC0-t | Up to 72 hours post last dose
  PK As Assessed By Area Under The Plasma Concentration Time Curve From Time 0 To The Time of The Last Quantifiable Concentration Of LP-168
PK Parameter AUC0-∞ | Up to 72 hours post last dose
  PK As Assessed By Area Under The Plasma Concentration Time Curve From Time 0 To The Time of Intersection of the extrapolated concentration-time curve and the time-axis Of LP-168 PK curve
PK Parameter Cmax | Up to 72 hours post last dose
  Pharmacokinetics (PK) As Assessed By Maximum Observed Plasma Concentration of LP-168
PK Parameter Tmax | Up to 72 hours post last dose
  PK As Assessed By Time To Maximum Observed Plasma Concentration of LP-168

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events as determined by CTCAE v5.0 | From the first dose of the study drug to 4 days after last dose]
Severity of Treatment Emergent Adverse Events as determined by CTCAE v5.0 | From the first dose of the study drug to 4 days after last dose]

CONTACTS AND LOCATIONS:
Overall Officials: Honggang Lou, MS, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No